CLINICAL TRIAL: NCT01497652
Title: A Double Blind Placebo Controlled Trial Evaluating Rasagiline Effects on Cognition in Parkinson's Disease Patients With Mild Cognitive Impairment Receiving Dopaminergic Therapy
Acronym: RECOGNIZE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Teva Neuroscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIT-TN-067
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Cognition; Rasagiline; MoCA; Mild Cognitive Impairment in Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Active Comparator): Treatment group will receive Rasagiline (Azilect) 1mg daily
  Interventions: Drug: Rasagiline
- Placebo Group (Placebo Comparator): will receive placebo daily
  Interventions: Drug: Rasagiline/Placebo

INTERVENTIONS:
Drug: Rasagiline/Placebo — Will receive placebo pills each day for the entire 14 weeks.
  Other Names: Sugar pill
  Arms: Placebo Group
Drug: Rasagiline — 0.5 mg for two weeks, then 1 mg for 12 weeks.
  Other Names: Azilect
  Arms: Treatment Group

SUMMARY:
The present pilot study is designed to assess the extent to which rasagiline may improve cognition in Parkinson's disease patients requiring dopaminergic therapy. The primary objective is to assess improvement in the Montreal Cognitive Assessment (MoCA) in patients who have been on rasagiline at 1mg daily for twelve weeks. The secondary objective is to assess changes in the SCOPA-COG, FAB, and UPDRS II & III at the end of week 14.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 40 or older with idiopathic Parkinson's disease on stable dopaminergic therapy for at least 1 month. The UK Brain Bank Criteria will be used to establish the diagnosis of Parkinson's disease. Women must be post menopausal or agree to avoid pregnancy. Modified Hoehn & Yahr staging < 3 and MoCA score must be greater than 21 but less than 28. Geriatric Depression Scale (GDS) is a sensitive and specific screen for depression in the Parkinson's disease population. GDS scores of < 5 will be included in the study.

Exclusion Criteria:

* Patients with secondary dementia, severe depression and atypical Parkinson's syndromes or Parkinson's plus will be excluded from the study. Patients on acetylcholine esterase or NMDA inhibitor medication will be excluded from the study. Patients with history of brain surgery for Parkinson's disease, stroke or significant head injury, active epilepsy will be excluded. Patients on Amantidine, neuroleptics, metoclopramide, alphamethyldopa within the last 6 months will be excluded. Individuals using meperidine, and tramadol will be excluded. Patients with congestive heart failure or myocardial infarction will also be excluded to avoid vascular dementia.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | 14 Weeks
  Best value is 30 and Worst Value is 0. Scores for a series of subscales are not combined for a total overall score.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando L Pagan, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States